CLINICAL TRIAL: NCT00780806
Title: An Open-Label Safety And Blood Collection Study In Mnb Rlp2086 Vaccinated Healthy Adult Volunteers For Immunological Assay Development
Brief Title: Safety And Blood Collection Study Of Meningococcal B Rlp2086 Vaccine In Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 6108A1-1003; B1971003
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Meningitis, Meningococcal
Keywords: MnB; rLP2086; blood collection; vaccination
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Immunization with one dose of MnB rLP2086 vaccine at 0, 1 and 6 months
  Interventions: Biological: meningococcal B rLP2086 vaccine candidate; Procedure: Blood draw

INTERVENTIONS:
Biological: meningococcal B rLP2086 vaccine candidate — vaccine, 0.5 mL, 3 doses, 0 - 2 - 6 to 9 months
Procedure: Blood draw — Blood draw

SUMMARY:
The purpose of this study is to evaluate the safety of an investigational meningococcal B rLP2086 vaccine in adults and to obtain blood samples from immunized subjects for use in assay development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject between the ages of >=18 and <=40 years
* Negative urine pregnancy test for all female subjects of childbearing potential prior to test article administration and at the completion of the study.
* All female or male subjects who are biologically capable of having children must agree to abstinence or commit to the use of a reliable method of birth control during for the duration of the study and for 30 days after early discontinuation. 4. Hemoglobin levels >=12.0 and <=16.5 g/dL for female subjects and >=13.0 and <=18.5 g/dL for male subjects.
* Blood pressure: Systolic blood pressure >90 and <160 mm Hg; Diastolic blood pressure >60 and <95 mm Hg.
* Body weight >=45 and <=120 kg.
* Able to be contacted by telephone during the study period.

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Prior vaccination with a serogroup B meningococcal vaccine.
* A previous anaphylactic or severe vaccine-associated adverse reaction.
* A known hypersensitivity to any study vaccine components.
* A known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids (excluding topical, inhalation and intra-articular corticosteroids).
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* Receipt of any blood products, including gamma globulin, in the period from 6 months before study vaccination through the study conclusion.
* Receipt of an inactivated vaccine within 14 days before study vaccinations and live attenuated vaccine within 28 days before study vaccination. This will apply throughout the study until the last vaccination.
* Any clinically significant chronic disease that, in the investigator's judgment may be worsened by blood draw.
* Received any investigational drug, vaccine or device within the 30-day period before study visit 1 and during the conduct of the study.
* History of culture-proven invasive disease caused by N meningitidis or N gonorrhoea.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety of 3 doses of MnB rLP2086 vaccine candidate assessed by frequency of solicited local and systemic reactions collected for 7 days after each study vaccination; evaluation of occurrence of AE and SAE during the duration of study | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Australia (3):
  - Pfizer Investigational Site, Herston
  - Pfizer Investigational Site, North Adelaide
  - Pfizer Investigational Site, Subiaco

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Marshall HS, Richmond PC, Nissen MD, Wouters A, Baber J, Jiang Q, Anderson AS, Jones TR, Harris SL, Jansen KU, Perez JL. A phase 2 open-label safety and immunogenicity study of a meningococcal B bivalent rLP2086 vaccine in healthy adults. Vaccine. 2013 Mar 15;31(12):1569-75. doi: 10.1016/j.vaccine.2013.01.021. Epub 2013 Jan 24. PMID 23352429
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6108A1-1003&StudyName=Safety%20And%20Blood%20Collection%20Study%20Of%20Meningococcal%20B%20Rlp2086%20Vaccine%20In%20Adults